## Effects Of Sensory Training and Electrical Stimulation on Sole of The Foot Sensations in Patients With Acute Hemiplegia

PT. CANSU HAYIROĞLU YEDITEPE UNIVERSITY 17.02.2020

## Informed Consent Form

This questionnaire is used within the scope of the research titled "Comparison of Footpad Sensory Training in Patients with Acute Hemiplegia and the Effect of Electrical Stimulation on Proprioceptive and Cortical Senses". The aim of this study is to compare the effects of neurodevelopmental physiotherapy program combined with sensory training or electrical stimulation on the sole of the foot in individuals diagnosed with hemiplegia. 30 patients diagnosed with acute hemiplegia will be included in the study, and physiotherapy sessions will take 20 minutes, with a total of 15 sessions 5 days a week.

You have to fill in the forms that we ask you to fill in the research correctly and notify us if you have any complaints or discomfort. We want you to know that you have the right to go out of the research at any time. There is no risk in the applications that will be applied within the scope of this research and no application will harm you. No fee is requested from you within this research. You will not be paid, as you are involved in this research. Your personal information will not be shared with corporate executives or third parties for any purpose.

Thank you for your participation.

Researcher: PT. Cansu HAYIROĞLU-+905378405948 (Person who can be reached 24 hours during the research)

I have read the information that should be given to the participant / volunteer in the study named Foot Base Sensory Training and the Effect of Electrical Stimulation on Proprioceptive and Cortical Senses in Patients with Acute Hemiplegia, and I fully understood the scope and purpose of the study I was asked to participate in, voluntarily. Written and verbal explanation about the study was made by the researcher named. I understood that I could quit this study whenever I wanted and without having to give any reason, and I would not face any negative if I quit.

In these circumstances, I agree to participate in this research voluntarily, without any pressure or coercion.

Volunteer's Name Surname / Signature / Date

Announcer's Name Surname / Signature / Date